CLINICAL TRIAL: NCT06906367
Title: A Prospective, Observational Study of Patients With Fabry Disease (US Specific)
Brief Title: A Study of Patients With Fabry Disease (US Specific)
Status: Recruiting | Type: Observational
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: AT1001-030X
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-03

CONDITIONS: Fabry Disease
Keywords: migalastat; AT1001; registry; lysosomal disease
MeSH Terms: conditions — Fabry Disease | interventions — migalastat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood, plasma, and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Migalastat-treated: Migalastat-treated patients at the time of enrollment who started the treatment within the 24 months prior to enrollment.
  Interventions: Drug: migalastat HCl
- ERT-treated: Patients receiving ERT at the time of enrollment who started the treatment within the 24 months prior to enrollment.
  Interventions: Drug: ERT
- Untreated: Untreated patients at the time of enrollment; these patients must never have been on therapy for Fabry disease prior to enrollment into the study and must meet criteria for receiving treatment with migalastat.

INTERVENTIONS:
Drug: migalastat HCl — Non-interventional study of participants receiving migalastat HCl 150 mg
  Groups: Migalastat-treated
Drug: ERT — Non-interventional study of participants receiving enzyme replacement therapy
  Groups: ERT-treated

SUMMARY:
This is an observational study to evaluate the effects of treatment on long-term effectiveness, safety, and health-related quality of life (HRQOL) in patients with Fabry disease, with a main focus on migalastat.

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational, effectiveness, safety, and outcomes study enrolling at least 450 patients with Fabry disease globally (at least 250 patients in the migalastat-treated group, approximately 100 patients in the ERT-treated group, and approximately 100 patients in the untreated group [patients who have never been on treatment for Fabry disease]). Enrollment will continue for a period of 5 years and all patients will be followed for up to 5 years after their enrollment.

Disclaimer: This is a global study, the country level requirements may vary from site to site. The requirements noted in this posting are specific to the US.

ELIGIBILITY:
I. Migalastat-treated patients (Commercial only participants)

1. Patients with Fabry disease 18 years or older with amenable GLA variants who have commenced commercial migalastat treatment within 24 months preceding enrollment, who have an eGFR greater than or equal to 30 mL/min/1.73 m2 at the time of enrollment and are still taking migalastat at the time of enrollment, or who are starting migalastat at the time of enrollment, excluding those who participated in a prior migalastat clinical trial
2. Patients who show a decline in their Fabry disease symptomatology based on any of the following:

   1. a decrease in annualized rate of decline eGFRCKD-EPI of ≥ 2 mL/min/1.73 m2 during the 2 years prior to enrollment
   2. microalbuminuria/macroalbuminuria (≥ 30 mg/24 h or ≥ 20 mg on first morning urine) or urine ACR of ≥ 30 mg/g (via spot urine collection) at any time prior to or at enrollment
   3. proteinuria (> 0.5 g/g UPCR) any time prior to or at enrollment
   4. males with classic Fabry disease phenotype

II. Migalastat-treated patients who are not considered to be in renal decline (Commercial migalastat users only)

1. Patients with Fabry disease with amenable GLA variants who have been on commercial migalastat regardless of the duration of treatment

III. Migalastat-treated patients (Prior clinical trial participants)

1. Patients with Fabry disease 18 years or older who had commenced treatment with migalastat while in a clinical trial and were exposed to treatment for at least 24 months preceding enrollment, who have an eGFR greater than or equal to 30 mL/min/1.73 m2 at the time of enrollment, and who are still taking migalastat at the time of enrollment, having switched to commercial product

IV. Untreated patients

1. Patients with Fabry disease 18 years or older with amenable GLA variants, who have never been on treatment for Fabry disease, who have an eGFR greater than or equal to 30 mL/min/1.73 m2 at the time of enrollment, and who meet local treatment guidelines for Fabry disease
2. Patients who show a decline in their Fabry disease symptomatology based on any of the following:

   1. a decrease in annualized rate of decline eGFRCKD-EPI of ≥ 2 mL/min/1.73 m2 during the 2 years prior to enrollment
   2. microalbuminuria/macroalbuminuria (≥ 30 mg/24 h or ≥ 20 mg on first morning urine) or urine ACR of ≥ 30 mg/g (via spot urine collection) at any time prior to or at enrollment
   3. proteinuria (> 0.5 g/g UPCR) any time prior to or at enrollment
   4. males with classic Fabry disease phenotype

V. ERT-treated patients

1. Patients with Fabry disease 18 years or older who have commenced ERT within 24 months preceding enrollment, who have an eGFR greater than or equal to 30 mL/min/1.73 m2 at the time of enrollment and are still being treated with ERT at the time of enrollment, and who have amenable GLA variants
2. Patients who show a decline in their Fabry disease symptomatology based on any of the following:

   1. a decrease in eGFRCKD-EPI annualized rate of decline of ≥ 2 mL/min/1.73 m2 during the 2 years prior to enrollment
   2. microalbuminuria/macroalbuminuria (≥ 30 mg/24 h or ≥ 20 mg on first morning urine) or urine ACR of ≥ 30 mg/g (via spot urine collection) at any time prior to or at enrollment
   3. proteinuria (> 0.5 g/g UPCR) any time prior to or at enrollment
   4. males with classic Fabry disease phenotype

All patients 1. All treated and untreated patients with Fabry disease who are enrolled in the study must be able to understand and provide written informed consent or assent.

Exclusion Criteria

1. Patients who currently are participating in a clinical trial of any investigational medicinal product or device at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Globally, approximately 450 patients with classic and late onset/nonclassic phenotypes of Fabry disease will be enrolled, with approximately 250 patients in the migalastat-treated group, 100 in the ERT-treated group, and approximately 100 patients in the untreated group.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2032-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of change in Estimated Glomerular Filtration Rate (eGFR) | Baseline and prospective up to 5 years
  Annualized rate of change in eGFR(CKD-EPI) over time from study enrollment for the comparison between migalastat-treated and untreated patients who have risk factors for eGFR decline

SECONDARY OUTCOMES:
Time to the first Fabry-associated clinical event (FACE) | Baseline and prospective up to 5 years
  Time to first FACE, which are cardiac, cerebrovascular, and renal events, and death due to FACEs, from enrollment in the study to compare between migalastat-treated and untreated patients.
Time to the first Fabry-associated clinical event (FACE) | Retrospective and prospective up to 5 years
  Time to first FACE, which are cardiac, cerebrovascular, and renal events, and death due to FACEs, from start of treatment to compare between migalastat-treated and ERT-treated patients.
Annualized rate of change in Estimated Glomerular Filtration Rate (eGFR) | Retrospective and prospective up to 5 years
  Annualized rate of change in eGFR(CKD-EPI) from start of treatment over time for the comparison between migalastat-treated and ERT-treated patients
Incidence and occurrence of FACE | Retrospective and prospective up to 5 years
  Incidence and occurrence of FACE will be evaluated overall, and separately by cardiac, cerebrovascular, and renal clinical events (including death in these categories)
Changes in plasma lyso Gb3 | Retrospective and prospective up to 5 years
  Biomarker of disease
Changes in WBC α-Gal A enzyme activity in males | Retrospective and prospective up to 5 years
  Biomarker of disease
Brief Pain Inventory (BPI)-Short Form | Baseline and prospective up to 5 years
  A 12-question form using a 10-point scale to allow patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function, along with a question about percentage of pain relief by analgesics
FABPRO-GI Short Form-v2-stomach pain domain | Baseline and prospective up to 5 years
  Three questions regarding GI signs and symptoms over a 7-day recall period and a Bristol Stool Scale (BSS), providing a pictorial chart and descriptive text for 7 types of stools. Using a 10-point scale, patients will rate the severity of their worst occurrence of stomach pain and diarrhea from 0 (none) to 10 (worst possible). Frequency and consistency of diarrhea will be assessed, as patients will provide the number of stools they have each day of BSS Type 1 through BSS Type 7.
FABPRO-GI Short Form-v2-diarrhea domain | Baseline and prospective up to 5 years
  Three questions regarding GI signs and symptoms over a 7-day recall period and a Bristol Stool Scale (BSS), providing a pictorial chart and descriptive text for 7 types of stools. Using a 10-point scale, patients will rate the severity of their worst occurrence of stomach pain and diarrhea from 0 (none) to 10 (worst possible). Frequency and consistency of diarrhea will be assessed, as patients will provide the number of stools they have each day of BSS Type 1 through BSS Type 7.
Weekly number of stools of BSS Types 6 and 7 (frequency) | Baseline and prospective up to 5 years
Number of days per week with at least 1 stool of BSS Type 6 or 7 (consistency) | Baseline and prospective up to 5 years
HRQOL by using PROs and health preference measures utility (SF-12) | Baseline and prospective up to 5 years
  Patient-reported health-related quality of life (HRQOL) will be assessed using Short Form-12 (SF-12): An abridged practical version of the 36-item Short Form Health Survey (SF-36), which contains 8 subscales: physical functioning (2 items), role limitations due to physical problems (2 items), bodily pain (1 item), general health perceptions (1 item), vitality (1 item), social functioning (1 item), role limitations due to emotional problems (2 items), and mental health (2 items)
HRQOL by using PROs and health preference measures utility (EQ-5D) | Baseline and prospective up to 5 years
  Patient-reported health-related quality of life (HRQOL) will be assessed using EuroQol-5D (EQ-5D), a preference-based HRQOL measure with 1 question for each of the 5 dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D questionnaire also includes a Visual Analog Scale, by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status)
HRQOL by using PROs and health preference measures utility (TSQM-9) | Baseline and prospective up to 5 years
  Patient-reported health-related quality of life (HRQOL) will be assessed using Treatment Satisfaction Questionnaire for Medications-9 (TSQM-9, migalastat-treated patients only): A generic measure of treatment satisfaction for medication which assesses patient perception of effectiveness, side effects, convenience, and global satisfaction
Occurrence of SAEs | Baseline and prospective up to 5 years
Overall survival among all patients enrolled | Baseline and prospective up to 5 years
  Assessed by recorded patient deaths from any cause
Number of participants with male infertility | Baseline and prospective up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research, Study Director — Amicus Therapeutics
Locations (7):
- United States (7):
  - UAB Nephrology Research Clinic at Paula Building, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Emory Genetics, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Renal Disease Research Institute, Dallas, Texas
  - Lysosomal and Rare Disorders Research and Treatment Center, Inc., Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing proposals and requests will be reviewed on a case-by-case basis. Requests for data should be addressed to Nick Rees at nrees@amicusrx.com. Requests will be reviewed by a medical steering committee.